CLINICAL TRIAL: NCT00528645
Title: Phase II Study of the c-SRC Inhibitor AZD0530 After Four Cycles of Cytoreductive Chemotherapy for Patients With Extensive Stage Small Cell Lung Carcinoma
Brief Title: AZD0530 in Treating Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01831; NCI-2012-01831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCTG-N0621; CDR0000563952; N0621 (Other: North Central Cancer Treatment Group); N0621 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Lung Metastases; Malignant Pleural Effusion; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Small Cell Lung Carcinoma | interventions — saracatinib

ARMS (1):
- Treatment (saracatinib) (Experimental): Patients receive oral AZD0530 once daily for up to 2 years in the absence of disease progression or unacceptable toxicity. Blood samples are obtained at baseline and periodically during study to determine levels of circulating tumor cells for defined translational studies.
  Interventions: Drug: saracatinib

INTERVENTIONS:
Drug: saracatinib — Given orally
  Other Names: AZD0530

SUMMARY:
AZD0530 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase II study is studying how well giving AZD0530 works in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 12-week progression-free survival rate of patients with extensive stage small cell lung cancer treated with AZD0530.

SECONDARY OBJECTIVES:

I. To determine the response rate in patients treated with this drug. II. To determine the overall survival and time-to-progression in patients treated with this drug.

III. To determine the adverse events of AZD0530 in these patients IV. To determine the effect of AZD0530 treatment on levels of circulating tumor cells in these patients.

V. To determine potential predictive markers of response in circulating tumor cells after treatment with this drug.

VI. To evaluate the rate of tumor marker (i.e., circulating tumor cells) stabilization in patients treated with this drug.

TERTIARY OBJECTIVES:

I. To determine the effect of AZD0530 treatment on levels of circulating tumor cells.

II. To determine potential predictive markers of response in circulating tumor cells after treatment with this drug.

III. To evaluate the rate of tumor marker (i.e., circulating tumor cells) stabilization in patients treated with this drug.

OUTLINE: Patients receive oral AZD0530 once daily for up to 2 years in the absence of disease progression or unacceptable toxicity. Blood samples are obtained at baseline and periodically during study to determine levels of circulating tumor cells for defined translational studies.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer

  * No mixed histology
* Extensive stage disease, defined as any of the following:

  * Metastatic disease outside the chest
  * Contralateral supraclavicular nodes or contralateral hilar nodes that cannot be included in a single radiation port
  * Cytologically confirmed malignant pleural effusion

    * Clinically significant effusions (e.g., symptomatic pleural effusion) must be drained prior to treatment
* Previously untreated disease* OR stable disease, partial response, or complete response ≤ 4 weeks after completion of one course (four 3-week courses) of standard platinum-based chemotherapy
* No symptomatic, untreated, or uncontrolled CNS metastases

  * CNS metastases previously treated with whole brain radiotherapy allowed
* ECOG performance status (PS) 0-2
* Life expectancy ≥ 12 weeks
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin > 9.0 g/dL
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* ALT and AST ≤ 3 times ULN (≤ 5 times ULN if liver involvement)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Proteinuria ≤ +1 on two consecutive dipsticks taken no less than 24hours apart
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective protection during and for up to 8 weeks after completion of study therapy
* QTc interval ≤ 460 msec
* No seizure disorder
* No significant traumatic injury ≤ 4 weeks prior to registration
* No clinically significant infection
* No HIV-positivity
* No second primary malignancy, except for carcinoma in situ of the cervix or nonmelanoma skin cancer, unless prior malignancy was diagnosed and treated ≥ 5 years with no subsequent evidence of recurrence

  * Patients with a history of low grade(Gleason score ≤ 6) localized prostate cancer will be eligible even if diagnosed < 5 years prior to registration
* No concurrent severe and/or uncontrolled medical conditions, including any of the following:

  * Cardiac arrhythmias
  * Angina pectoris uncontrolled with medication
  * Myocardial infarction within the past 3 months
  * Significant ECG abnormalities
  * Hypertension, labile hypertension, or history of poor compliance with anti-hypertensive medication
  * Congestive heart failure within the past 3 months, unless ejection fraction > 40%
  * Interstitial pneumonia or extensive, symptomatic interstitial fibrosis of the lung
  * Poorly controlled diabetes
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to AZD0530
* No condition that impairs the ability to swallow AZD0530 tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or requiring IV alimentation
  * Prior surgical procedures affecting absorption of AZD0530 tablets
  * Active peptic ulcer disease
* No serious condition that, in the opinion of the investigator, would compromise the patient's ability to complete the study
* At least 4 weeks since prior major surgery (i.e., laparotomy) or open biopsy
* At least 2 weeks since prior minor surgery
* At least 4 weeks since any prior investigational ancillary therapy (i.e., utilized for a non-FDA-approved indication and in the context of a research investigation)
* At least 7 days since prior use of strong inhibitors of CYP3A4 and no concurrent use for up to 7 days after discontinuation of AZD0530
* Prior nonthoracic palliative radiotherapy allowed
* Concurrent bisphosphonates for treatment of lytic metastatic bone disease allowed at the discretion of the treating physician
* No concurrent prophylactic granulocyte colony-stimulating factor (i.e., G-CSF)
* No concurrent products that stimulate thrombopoiesis
* No concurrent St. John's wort
* No other concurrent chemotherapy, immunotherapy, hormonal therapy,or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 patients were enrolled from 13 medical clinics from February 5, 2008 to August 21, 2008.
Pre-assignment Details: One patient cancelled prior to treatment initiation and is excluded in the analysis.
Groups:
- Treatment (Saracatinib): Patients receive oral AZD0530 once daily for up to 2 years in the absence of disease progression or unacceptable toxicity.
  saracatinib : saracatinib 175mg given orally daily with re-treatment every 3 weeks
Period: Overall Study
Arm/Group | Treatment (Saracatinib)
Started | 23
Completed | 20
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Saracatinib): Patients receive oral AZD0530 once daily for up to 2 years in the absence of disease progression or unacceptable toxicity. Blood samples are obtained at baseline and periodically during study to determine levels of circulating tumor cells for defined translational studies.
  saracatinib : saracatinib 175mg given orally daily with re-treatment every 3 weeks
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 58 [48 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 12 Weeks
Description: The progression-free survival (PFS) rate at 12 weeks will be estimated by calculating the number of patients that are alive and progression-free at 12 weeks post-registration divided by the total number of evaluable patients and multiplied by 100. All patients meeting the eligibility criteria who have signed a consent form, begun AZD0530 treatment, and are not lost to follow-up before 12 weeks, will be considered evaluable for the 12-week progression-free survival (PFS) rate.
  Progression is defined using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progression is defined as having a new lesion or having at least a 20% increase in the sum of the longest diameter of target lesions from baseline.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Saracatinib): Patients receive oral AZD0530 once daily for up to 2 years in the absence of disease progression or unacceptable toxicity.
  saracatinib: saracatinib 175mg given orally daily with re-treatment every 3 weeks
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 23
percentage of participants | 26 [10 to 48]

2. Secondary Outcome: Overall Survival
Description: Overall Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment (Saracatinib): saracatinib : saracatinib 175mg given orally daily with re-treatment every 3 weeks
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 23
months | 7.8 [6.9 to 10.6]

3. Secondary Outcome: Confirmed Tumor Response (Defined as Complete or Partial Response on 2 Consecutive Evaluations at Least 4 Weeks Apart)
Description: Response was assessed using the RECIST v1.1 criteria. Patients were evaluated after every other cycle (after cycle 2, 4, 6, etc...) and when progression is suspected. A Complete Response (CR) is defined as the disappearance of all target lesions. A Partial Response (PR) is defined as at least a 20% decrease in the sum of the longest diameter of target lesions from baseline. A confirmed response is defined as a CR or PR as the objective status on 2 consecutive evaluations at least 4 weeks apart..
Time Frame: After every other 21-day cycle, up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 23
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0

4. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) is defined as the time from registration to documentation of disease progression or death, whichever occurs first. The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to documentation of disease progression or death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 23
months | 1.5 [1.3 to 1.6]

ADVERSE EVENTS:
Arm/Group | Treatment (Saracatinib)
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=23)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=23)
Hemoglobin decreased (Blood and lymphatic system disorders) | 20 (39)
Diarrhea (Gastrointestinal disorders) | 6 (26)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (12)
Vomiting (Gastrointestinal disorders) | 7 (9)
Fatigue (General disorders) | 16 (45)
Fever (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 8 (19)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 7 (8)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Headache (Nervous system disorders) | 2 (2)
Taste alteration (Nervous system disorders) | 2 (2)
Protein urine positive (Renal and urinary disorders) | 6 (18)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (6)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less